CLINICAL TRIAL: NCT07134582
Title: The Effects of Hippotherapy on Viscoelastic Properties of Thoracolumbar Fascia and Quality of Life in Children With Spastic Cerebral Palsy and Their Parents/Caregivers
Brief Title: Trial Examines Short-term Effects of Hippotherapy on Fascia Properties and Quality of Life in Children With CP.
Acronym: HYPPOTER25
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HYPPOTER25
Record Dates: First submitted 2025-07-31; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy (CP); Rehabilitation; Motor Coordination or Function; Hippotherapy; Fascia; Quality of Life
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hippotherapy 1x/week (Experimental)
  Interventions: Other: Hippotherapy 1x/week
- Hippotherapy 2x/week (Experimental)
  Interventions: Other: Hippotherapy 2x/week
- Control (No Intervention)

INTERVENTIONS:
Other: Hippotherapy 1x/week — This group will perform hippotherapy once per week for 12 weeks
  Arms: Hippotherapy 1x/week
Other: Hippotherapy 2x/week — This group will perform hippotherapy twice per week for 12 weeks
  Arms: Hippotherapy 2x/week

SUMMARY:
The effects of hippotherapy on gross motor function, balance, and spasticity in children with cerebral palsy (CP) are well-documented, but its impact on the thoracolumbar fascia (TLF) remains unexplored area to date. This research protocol aims to investigate the short-term effects of hippotherapy on the viscoelastic and biomechanical properties of the TLF and quality of life (QoL) in children with spastic CP and their parents/caregivers. A 4-week randomized control trial will compare the effects of once-weekly and twice-weekly hippotherapy sessions to a control group without intervention. The study will assess the viscoelastic and biomechanical properties of the TLF using the MyotonPRO device in children with spastic CP aged 4-12 years. Myotonometer parameters, including oscillation frequency, stiffness, logarithmic decrement, stress relaxation, and creep, will be analyzed before, during, and after the intervention. Functional tests, such as the 10-meter walk test (comfortable and fast walking), cadence, one-leg stance test (eyes open and closed), and functional reach test (forward and lateral), will also be monitored. QoL will be assessed using the CP QOL-Child questionnaire. The primary outcomes will include changes in myotonometer parameters, their correlation with functional tests, and differences between intervention groups. Secondary outcomes will explore whether hippotherapy impacts QoL and the relationship between QoL domains and TLF properties. Results will evaluate whether twice-weekly therapy yields statistically significant differences in the specified parameters compared once-weekly sessions and contribute to understanding hippotherapy's mechanisms, supporting more individualized therapies to improve QoL for children with CP and their families.

ELIGIBILITY:
Inclusion Criteria:

* classified as level II or III according to the GMFCS, and who, according to the assessment of a specialist physician, are indicated for hippotherapy aged between 4 and 12 years
* who are undergoing neurophysiotherapeutic treatment
* who have not undergone orthopedic surgery in the last six months and do not have uncontrolled epilepsy
* are willing to be randomly assigned to any group (or whose parents/caregiver's consent)
* understand instructions in Slovene and are willing to participate in the study for four weeks (or whose parents/ caregiver's consent)
* without skin diseases, scars, or wounds on the examined part of the back

Exclusion Criteria:

* who have previously participated in a hippotherapy program
* with a known and diagnosed psychiatric disorder for which hippotherapy is contraindicated
* with limitations due to hearing or visual impairment
* with painful adductor contractures, painful subluxation, or hip dislocation are not willing to be randomly assigned to any group (or whose parents/caregiver's consent)
* who are afraid of horses or have an allergy to horsehair
* with skin diseases, scars, or wounds on the examined part of the back

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in viscoelastic properties in TLF (5 measurable parameters) | 1. baseline (before hippotherapy starts): all groups 2. in 2 weeks (midway through the therapy): all groups 3. in 4 weeks (at the end of hippotherapy): all groups 4. one day after the completion of the 4-week hippotherapy: only experimental groups
  1. oscillation frequency (F)-Hz
  2. dynamic stiffness (S)-N/m
  3. oscillation decrement (D)-arb
  4. mechanical stress relaxation time (R)-ms (milliseconds)
  5. creep (C)-arb
Functional tests (7 measurable parameters) | 1. baseline (before hippotherapy starts): all groups 2. in 2 weeks (midway through the therapy): all groups 3. in 4 weeks (at the end of hippotherapy): all groups 4. one day after the completion of the 4-week hippotherapy: only experimental groups
  1. 10-meter walk test (comfortable walking)-10 m/time spent in seconds
  2. 10-meter walk test ( fast walking)-10 m/time spent in seconds
  3. cadence (steps/minute)
  4. a one-leg stance test with eyes open-seconds
  5. a one-leg stance test with eyes closed-seconds
  6. functional reach test forward-centimetres
  7. functional reach test lateral-centimetres

SECONDARY OUTCOMES:
Quality of life of children and Quality of live of their parents/caregivers | 1. baseline (before hippotherapy starts) 2. in 4 weeks (at the end of hippotherapy)
  CP QOL-Child questionnaire (version for children) to children aged between 9 and 12 years in both experimental groups.
  CP QOL-Child questionnaire (version for parents) to the parents/caregivers of all children in both experimental groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Konjeniški zavod Epona, Novo Mesto, Dolenjska, Slovenia

IPD SHARING:
Plan to Share IPD: No